CLINICAL TRIAL: NCT03479918
Title: Randomized, Controlled (Comparative), Open, Prospective Study Evaluating an Efficacy of R-DA-EPOCH-21, R-BL-M-04 and Autologous Stem Cells Transplantation in Patients With High-Grade B-cell Lymphoma Double-hit and High-Grade B-cell Lymphoma Not Otherwise Specified
Brief Title: R-BL-M-04 Versus R-(DA)-EPOCH and Autologous Stem Cells Transplantation in Patients With High-Grade B-cell Lymphoma Double-hit (HGBL DH) and High-Grade B-cell Lymphoma Not Otherwise Specified (HGBL NOS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elena N.Parovichnikova (Network)
Responsible Party: Sponsor-Investigator, Elena N.Parovichnikova, Head of BMT department, National Research Center for Hematology, Russia, National Research Center for Hematology, Russia
Organization: National Research Center for Hematology, Russia (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGBL DH and HGBL NOS
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma, High-Grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R-DA-EPOCH-21 (Active Comparator): The protocol involves 4-6 cycles. Intrathecal administration of dexamethasone 4 mg, methotrexate 15 mg and cytarabine 30 mg is required once during chemotherapy. In case of CNS involvement intrathecal administration is repeated 3 times a week till the normal cell count in cerebrospinal liquid.
  Interventions: Drug: R-DA-EPOCH-21
- R-BL-M-04 (Active Comparator): Course A:
  Rituximab 375 mg/m2 IV 0 day, Dexamethasone 10 mg/m2/day IV 1 - 5 days, Methotrexate 1500 mg/m2 12 h IV 1 day, Ifosfamide 800 mg/m2/day 1 h IV 1 - 5 days, Etoposide 100 mg/m2/day IV 4, 5 days, Doxorubicin 50 mg/m2/day IV day 3, Vincristine 2 mg IV 1 day, Cytarabine 150 mg/m2/day IV 1 h 4, 5 days.
  Course C:
  Rituximab 375 mg/m2 IV 0 day, Dexamethasone 10 mg/m2/day IV 1 - 5 days, Methotrexate 1500 mg/m2 12 h IV 1 day, Vinblastine 5 mg/m2 IV day 1, Cytarabine 2000 mg/m2/day IV 3 h 2, 3 days, Etoposide 150 mg/m2/day IV 3-5 days.
  Intrathecal administration of dexamethasone 4 mg, methotrexate 15 mg and cytarabine 30 mg is required once during chemotherapy. In case of CNS involvement intrathecal administration is repeated 3 times a week till the normal cell count in cerebrospinal liquid.
  Interventions: Drug: R-BL-M-04
- R-DA-EPOCH-21 + auto-SCT (Active Comparator): The protocol involves 4-6 cycles. Patients with complete remission after 4 cycles undergo auto-SCT.
  Intrathecal administration of dexamethasone 4 mg, methotrexate 15 mg and cytarabine 30 mg is required once during chemotherapy. In case of CNS involvement intrathecal administration is repeated 3 times a week till the normal cell count in cerebrospinal liquid.
  Interventions: Drug: R-DA-EPOCH-21 + auto-SCT
- R-BL-M-04 + auto-SCT (Active Comparator): The protocol involves 4 cycles. Patients with complete remission after 4 cycles undergo auto-SCT.
  Intrathecal administration of dexamethasone 4 mg, methotrexate 15 mg and cytarabine 30 mg is required once during chemotherapy. In case of CNS involvement intrathecal administration is repeated 3 times a week till the normal cell count in cerebrospinal liquid.
  Interventions: Drug: R-BL-M-04 + auto-SCT

INTERVENTIONS:
Drug: R-DA-EPOCH-21 — R-DA-EPOCH-21 treatment without auto-SCT for HGBL DH and HGBL NOS patients younger than 60 years. Courses are repeated every 21 days.
  Other Names: R-DA-EPOCH
  Arms: R-DA-EPOCH-21
Drug: R-BL-M-04 — R-BL-M-04 treatment without auto-SCT for HGBL DH and HGBL NOS patients younger than 60 years. Courses are repeated every 21 days.
  Arms: R-BL-M-04
Drug: R-DA-EPOCH-21 + auto-SCT — R-DA-EPOCH-21 treatment with auto-SCT for HGBL DH and HGBL NOS patients younger than 60 years. Courses are repeated every 21 days.
  Other Names: R-DA-EPOCH + auto-SCT
  Arms: R-DA-EPOCH-21 + auto-SCT
Drug: R-BL-M-04 + auto-SCT — R-BL-M-04 treatment with auto-SCT for HGBL DH and HGBL NOS patients younger than 60 years. Courses are repeated every 21 days.
  Arms: R-BL-M-04 + auto-SCT

SUMMARY:
Purpose: to evaluate an efficacy of chemotherapy regimens R-DA-EPOCH-21 and R-BL-04 with and without autologous hematopoietic stem cells transplantation (auto-SCT) in newly diagnosed patients with High-Grade B-cell Lymphoma Double-hit and High-Grade B-cell Lymphoma Not Otherwise Specified.

DETAILED DESCRIPTION:
Patients initially are randomized into 4 arms:

the first arm R-DA-EPOCH-21 the second arm R-BL-M-04 the third arm R-DA-EPOCH-21 + auto-SCT the fourth arm of R-BL-M-04 + auto-SCT Patients who achieved complete remission after 6 cycles of R-DA-EPOCH-21 or 4 cycles of R-BL-M-04 immunochemotherapy continue to be under observation (1st and 2nd arms) or continue treatment with Rituximab + BCNU+Etoposid+Ara-C+Melphalan (R-BEAM) followed by auto-SCT (3rd and 4th arms).

Patients who did not achieve complete remission with PET-CT data (4-5 Deauville points) are removed from the protocol and undergoing second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. First established the diagnosis of HGBL DH or HGBL-NOS.
2. No previous treatment with chemotherapy and/or radiation therapy of DLBCL
3. Informed consent of the patient.

Exclusion Criteria:

1. Pretreated lymphoma.
2. HIV-associated lymphoma
3. Congestive heart failure, unstable angina, severe cardiac arrhythmias and conduction disturbances, myocardial infarction.
4. Renal insufficiency (serum creatinine greater than 0.2 mmol/L) (except cases with specific kidney infiltration, urinary tract compression by tumour conglomerate or presence of uric acid nephropathy due to massive cytolysis syndrome).
5. Liver failure (except cases with liver tumour infiltration), acute hepatitis or active phase of chronic hepatitis B or C with serum bilirubin greater than 1.5 standards, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 3 standards, prothrombin index less than 70%.
6. Severe pneumonia (except cases with specific lungs infiltration), accompanied by respiratory failure (dyspnea > 30 in min., hypoxemia less than 70 mm Hg, when it is impossible to compensate situation in 2-3 days).
7. Life-threatening bleeding (gastrointestinal, intracranial), with exception of bleeding due to tumour infiltration of organs (stomach, intestines, uterus, etc.) and disseminated intravascular coagulation due to underlying disease complications after their successful conservative treatment.
8. Severe mental disorders (delusions, severe depressive syndrome and other manifestations of productive symptoms) not related to specific infiltration of a central nervous system.
9. Decompensated diabetes.

11. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival
Relapse-free survival | 2 years
  Relapse-free survival
Progression | 2 years
  Frequency of progression

SECONDARY OUTCOMES:
Complete remission | 1 year
  Frequency of complete remission
Partial remission | 1 year
  Frequency of partial remission

OTHER OUTCOMES:
Probability of relapse or progression | 2 years
  Probability of relapse or progression

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnokva, PhD, Principal Investigator — National Research Center for Hematology, Moscow, Russian Federation
Locations (1):
- National Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No